CLINICAL TRIAL: NCT03535662
Title: A Phase 1, Open-Label, Single-Sequence Crossover Study in Healthy Male Participants to Determine the Effect of an Inhibitor of Cytochrome P450 3A and P Glycoprotein on Exposure to Orvepitant
Brief Title: A Pharmacokinetic Study of the Effect of Itraconazole Exposure to Orvepitant in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nerre Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ORV-1-01
Record Dates: First submitted 2018-05-11; First posted 2018-05-24 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Pharmacokinetic Study in Healthy Male Volunteers
MeSH Terms: interventions — orvepitant; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Orvepitant (Experimental): Orvepitant single 20mg dose
  Interventions: Drug: Orvepitant
- Orvepitant and itraconazole (Experimental): Orvepitant single 20mg dose in combination with repeat dose itraconazole
  Interventions: Drug: Orvepitant; Drug: Itraconazole

INTERVENTIONS:
Drug: Orvepitant — Single oral dose
Drug: Itraconazole — Once daily dosing for 10 days
  Arms: Orvepitant and itraconazole

SUMMARY:
A Phase 1 study to assess the effect of itraconazole, a strong inhibitor of CYP3A and P-glycoprotein, on the pharmacokinetics (PK) of orvepitant in healthy male volunteers.

Subjects will receive two single doses of 20mg orvepitant, once alone and once in combination with repeat doses of itraconazole. All subjects will follow the same sequence - orvepitant alone followed by orvepitant in combination with itraconazole.

ELIGIBILITY:
Key Inclusion Criteria:

* male volunteers
* judged to be in good health, based on the results of medical history, physical examination, vital signs, 12 lead ECG, and clinical laboratory findings
* body weight greater than 50 kg and body mass index (BMI) within the range 18 to 30 kg/m2 (inclusive)

Key Exclusion Criteria:

* clinically significant findings on physical examination
* relevant medical history
* history of or considered at high risk of seizures (except febrile fits in childhood), including history of significant head injury
* positive serology for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (anti-HCV) or human immunodeficiency virus (HIV)
* serum biochemistry and full blood count considered by the Investigator to be of clinical significance
* systolic blood pressure <100 or >140 mmHg or diastolic BP <50 or ˃90 mmHg, measured prior to the first dose of orvepitant
* abnormal 12 lead electrocardiogram (ECG)
* has donated one or more units (approximately 450 mL) of blood or acute loss of an equivalent amount of blood within 90 days prior to study intervention administration

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-09 (Actual)

PRIMARY OUTCOMES:
Exposure to orvepitant | 0 to 168 hours post dose
  Area Under Curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — PAREXEL EPCU
Locations (1):
- Parexel Epcu, Harrow, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No